CLINICAL TRIAL: NCT02613468
Title: A Comparative Evaluation in Pregnant Women of the Periodontal Condition and Low Birth Delivery Incidence
Brief Title: Periodontal Condition in Pregnancy and Low Birth Delivery Incidence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, İnci Devrim, Principal Investigator, Ondokuz Mayıs University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: OndokusMu
Record Dates: First submitted 2015-11-13; First posted 2015-11-24 (Estimated); Last update posted 2015-11-25 (Estimated); Status verified 2015-11

CONDITIONS: Pregnancy; Birth Weight; Periodontal Diseases
Keywords: Pregnancy; Low birth weight; Gingivitis; Inflammation; Periodontitis
MeSH Terms: conditions — Birth Weight; Periodontal Diseases; Gingivitis; Inflammation; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Periodontally healthy (Placebo Comparator): Some periodontal measurements (attachment level, probing depth, gingival index, plaque index, and bleeding on probing) were performed in periodontally healthy pregnant. These measurements were performed at the end of each trimester.
  Parameters such as number of pregnancies, previous low birth weight, prenatal care, genital tract infection, use of antibiotics, smoking, tooth brushing habit and birth weight were evaluated.
  Intervation: Collection of periodontal records and pregnancy parameters.
  Interventions: Other: collection of periodontal records; Other: pregnancy parameters
- Periodontally diseased, untreated (Placebo Comparator): This group is comprised of individuals who do not accept treatment Some periodontal measurements (attachment level, probing depth, gingival index, plaque index, and bleeding on probing) were performed in periodontally healthy pregnant. These measurements were performed at the end of each trimester.
  Parameters such as number of pregnancies, previous low birth weight, prenatal care, genital tract infection, use of antibiotics, smoking, tooth brushing habit were evaluated.
  Birth weight was recorded at the end of pregnancy.
  Interventions: Other: collection of periodontal records; Other: pregnancy parameters
- Periodontally diseased, treated (Active Comparator): This group is comprised of individuals who agree to treatment. Some periodontal measurements (attachment level, probing depth, gingival index, plaque index, and bleeding on probing) were performed in periodontally healthy pregnant. These measurements were performed at the end of each trimester.
  Parameters such as number of pregnancies, previous low birth weight, prenatal care, genital tract infection, use of antibiotics, smoking, tooth brushing habit were evaluated.
  Initial Periodontal Therapy is completed (calculus elimination, root planning, polishing etc.) This treatment is considered to be the safest time for pregnant mothers was performed in 2 trimester.
  Birth weight was recorded at the end of pregnancy. Intervation: Collection of periodontal records and pregnancy parameters.
  Interventions: Other: collection of periodontal records; Other: pregnancy parameters; Other: Initial Periodontal Therapy

INTERVENTIONS:
Other: collection of periodontal records — 1. Clinic attachment level
  2. Probing depth
  3. Gingival index
  4. Plaque index
  5. Bleeding on probing were performed in all groups. These measurements were performed at the end of each trimester.
Other: pregnancy parameters — Parameters such as number of pregnancies, previous low birth weight, prenatal care, genital tract infection, use of antibiotics, smoking, tooth brushing habit and birth weight were evaluated.
Other: Initial Periodontal Therapy — Initial Periodontal Therapy is completed ( Supragingival and subgingival calculus elimination, root planning, polishing etc.) This treatment is considered to be the safest time for pregnant mothers was performed in 2 trimester.
  Arms: Periodontally diseased, treated

SUMMARY:
The objective of this study was the evaluation of periodontal condition in pregnant women and the effect of the treatment of periodontal disease upon low birth weight.

DETAILED DESCRIPTION:
This research was carried out in the following three centers: Samsun Birth and Children's Hospital, Department of Obstetrics and Gynecology of the Faculty of Medicine and Faculty of Dentistry of the University of Ondokuz Mayıs. 269 women in their first trimester were included in this study. Their ages ranged from 18-35 years, their height was above 150 cm and they have no history of any systemic disease. At the end of each trimester these measurements were performed: attachment level, probing depth, gingival index, plaque index, and bleeding on probing. According to the periodontal diagnosis the research population was divided into three groups: periodontally healthy women; periodontally diseased women, however rejection of treatment; periodontally diseased women, however acceptance of treatment.In this study one-way ANOVA, chi-square, conditional logistic regression analyses were used.

ELIGIBILITY:
Inclusion Criteria:

* Age:18-35 years
* Sure of her dates

Exclusion Criteria:

* systemic diseases (i.e., diabetes mellitus, cancer, hypertension, urolithiasis, parathyroid disease, diseases that compromise pregnancy)
* Less than two pregnancy

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 269 (Actual)
Dates: Start 2004-01; Primary Completion 2004-12 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Number of pregnancies | At 9th months
  Number of pregnancies (numbers)
Birth weight | At 9th months
  Birth weight (kg)

SECONDARY OUTCOMES:
Probing pocket depth | average of 2nd months, 5th months and 8th months
  The changes in probing pocket depth in time frame.Probing pocket depth was measured for determining severity of disease and clinic outcome.
Clinical attachment level | average of 2nd months, 5th months and 8th months
  The changes in clinical attachment level in time frame. Clinical attachment level was measured for determining severity of disease and clinic outcome.
Gingival index | average of 2nd months, 5th months and 8th months
  The changes in gingival index in time frame. Gingival index was recorded for classifying and evaluating (coronally) gingival inflammation.
Plaque index | average of 2nd months, 5th months and 8th months
  The changes in plaque index in time frame. Plaque index was recorded for determining and classifying oral hygiene status.
Bleeding on probing | average of 2nd months, 5th months and 8th months
  The changes in bleeding on probing in time frame. Bleeding on probing was recorded for classifying and evaluating (apically) gingival inflammation.